CLINICAL TRIAL: NCT05711966
Title: Comparison of "IN-REC-SUR-E" and LISA in Preterm Neonates With Respiratory Distress Syndrome: a Randomized Controlled Trial (IN-REC-LISA Trial)
Brief Title: Comparison of INRECSURE and LISA in Preterm Neonates With RDS
Acronym: INRECLISA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Dr. Behcet Uz Children's Hospital (Other); Universitair Ziekenhuis Brussel (Other); University of Melbourne (Other); University of California, San Diego (Other); University Hospital Schleswig-Holstein (Other); Shengjing Hospital (Other); Policlinico Casilino ASL RMB (Other); The University of Western Australia (Other); Catholic University of the Sacred Heart (Other); Maggiore Hospital Carlo Alberto Pizzardi (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Ospedali Riuniti Ancona (Other); Careggi Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Monash University (Other); S.Eugenio Hospital (Other); Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, VENTO GIOVANNI, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4933
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
Keywords: Respiratory Distress Syndrome; Surfactant; INRECSURE; LISA
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia | interventions — Ventilators, Mechanical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-REC-SUR-E (Experimental): INRECSURE infants will receive preintubation medications and HFOV starting at MAP 8 cmH2O; frequency 15 Hz, with volume-guarantee (1.5-1.7 mL/kg). The I:E will be 1:1. An oxygenation guid-ed lung recruitment procedure will be performed using stepwise increments then decrements in MAP. The starting MAP will be increased stepwise as long as SpO2 improves reducing the FiO2 keeping SpO2 within the target range (90-94 %) until the oxygenation no longer improves or the FiO2 is equal to or less than 0.25 (opening MAP). Next, the MAP will be reduced stepwise until the SpO2 deterio-rates (closing MAP). After a second recruitment maneuver at the opening pressure, the optimal MAP will be set 2 cmH2O above the closing MAP. Then 200 mg/kg of poractant alfa (Chiesi Farmaceutici S.p.A., Parma, Italy) via a closed administration system will administrate. Infants with sufficient res-piratory drive will be extubated within 30 minutes after surfactant administration starting nCPAP (7-9 cm H2O) or NIPPV.
  Interventions: Device: Ventilator for High-frequency Oscillatory Ventilation (HFOV)
- Less Invasive Surfactant Administration (Active Comparator): By contrast, infants allocated to the LISA group will receive 200 mg/kg of poractant alfa (Chiesi Farmaceutici S.p.A., Parma, Italy) according to the following protocol: during nasal CPAP with a pressure of 7-8 cm H2O, surfactant will be administered over 0.5-3 min using the SurfCath™ tracheal instillation catheter (VYGON S.A. - Ecouen, France), or a 4- 6 F end-hole catheter, according to local protocols. After the same pre-procedural medications, the catheters will be positioned during laryngoscopy with or without Magill forceps. The catheter will be connected to a syringe pre-filled with the surfactant, and the surfactant is instilled slowly. The infant's mouth will be closed. In cases of apnoea or bradycardia, positive pressure ventilation will be performed until recovery. After surfactant administration, CPAP (7-9 cm H2O) therapy (16) or NIPPV will be continued.
  Interventions: Device: Less invasive surfactant administration (LISA)

INTERVENTIONS:
Device: Ventilator for High-frequency Oscillatory Ventilation (HFOV) — This device will be used to perform an HFOV recruitment maneuver before surfactant administration
  Arms: IN-REC-SUR-E
Device: Less invasive surfactant administration (LISA) — SurfCath™ tracheal instillation catheter, or a 4- 6 F end-hole catheter, according to local protocols will be used for surfactant administration
  Arms: Less Invasive Surfactant Administration

SUMMARY:
The primary hypothesis of this study is that surfactant administration by INtubate-RECruit-SURfactant-Extubate (IN-REC-SUR-E), via a high frequency oscillatory ventilation recruitment maneuver increases survival without BPD at 36 weeks' gestational age in spontaneously breathing infants born at 24+0-27+6 weeks' gestation affected by Respiratory Distress Syndrome (RDS) and failing nasal CPAP or nasal intermittent positive pressure ventilation (NIPPV) during the first 24 hours of life compared to less invasive surfactant administration (LISA).

DETAILED DESCRIPTION:
BACKGROUND: RDS represents the main cause of respiratory failure in preterm infants and one of the major causes of perinatal morbidity and mortality. Surfactant is a well-established therapy in neonatology, but its optimal administration method remains unresolved, especially with the focus on avoiding MV in preterm infants born before 28 weeks' gestational age (i.e. extremely low gestational age newborns - ELGAN). Duration of MV is a key determinant of the se-verity of bronchopulmo-nary dysplasia (BPD). Although attractive and beneficial in clinical practice, the INtubate, SURfac-tant, Extubate (IN-SUR-E) method cannot be universally applied to all pre-term neonates due to non-homogeneous surfactant distribution and lung derecruitment during intu-bation, resulting in failure rate in preterm infants ranging from 19 % to 69 %. A recent randomized clinical trial showed that the application of a recruitment manoeuvre just before surfactant admin-istration, followed by rapid extubation (INtubate-RECruit-SURfactant-Extubate [IN-REC-SUR-E]), decreased the need for MV during the first 72 h of life compared with IN-SUR-E technique in ELGAN, without in-creasing the risk of adverse neonatal outcomes. Recent-ly, a less invasive surfactant administration (LISA) method was developed with surfactant intro-duced into the trachea of infants breathing spontaneously using a small catheter instead of an endo-tracheal tube. The LISA technique poten-tially combines the benefits of early surfactant treatment CPAP avoiding MV. The last network me-ta-analyses on the comparative efficacy of methods for surfactant administration found that among preterm infants, LISA technique was associated with lower likelihood of mortality, need for MV and BPD compared with IN-SUR-E, but these findings did not include comparison to IN-REC-SUR-E method. More importantly, data for ELGAN are not as robust as for the higher gestation age groups. The same Authors of meta-analysis agree that data for ELGAN are not as ro-bust as for higher gestation age group and that lung recruitment before sur-factant administration (IN-REC-SUR-E) represents a promising novel alternative. The investigators therefore de-signed this study to compare the IN-REC-SUR-E technique with LISA for evaluating the compara-tive effectiveness of these techniques in increasing the survival without BPD of ELGANs.

METHODS: The primary hypothesis of this study is that IN-REC-SUR-E via a HFOV recruitment maneuver increases survival without BPD at 36 weeks' gestational age in spontaneously breathing ELGAN and failing nCPAP or nasal intermittent positive pressure ventilation (NIPPV) during the first 24 hours of life compared to LISA treatment.

Study design: this study is an unblinded multi-center randomized trial of IN-REC-SUR-E vs. LISA in ELGANs.

Randomisation and Masking: infants will be allocated to one of the two treatment groups (1:1) ac-cording to a restricted randomization procedure. Stratification factors will include centre and gesta-tional age (24+0 to 25+6 weeks or 26+0 to 27+6 weeks). The table of allocation will not be disclosed to ensure concealment and the randomization will be provided through Research Electron-ic Data Capture (RedCap) web application. The assignment to intervention will be unmasked to all trial par-ticipants: parents, research staff, and medical team will be only aware of study group as-signment af-ter randomization procedures.

Management in the Delivery Room: Neonates will be stabilized after birth with positive pressure us-ing a neonatal mask and a T-piece system (i.e. Neopuff Infant Resuscitator ®, Fisher and Paykel, Auckland, New Zealand). All neonates will be started on nCPAP of at least 6 cm H2O via mask or nasal prongs. Newborns who do not breathe or who are persistently bradycardic within the first 60 seconds after birth will receive positive-pressure ventilation with initial FiO2 of 0.30. Infants that will be transitioned successfully to spontaneous breathing will be transferred to NICU on nCPAP (6-7 cm H2O) or NIPPV. The decision to intubate and start MV in the delivery room will be in ac-cordance with the American Heart Association Guidelines. Method and timing of umbilical cord clamping will be as per standard practice at each site.

Surfactant treatment Nasal CPAP or NIPPV in the NICU will perform by nasal prongs or nasal mask, with a pressure of 7-8 cm H2O or with a setting of peak inspiratory pressure of 12-15 cmH2O, positive end-expiratory pressure of 7-8 cmH2O and rate of 30-40 breaths/min, respectively. Infants will receive surfactant with IN-REC-SUR-E or LISA if they need a FiO2 ≥ 0.30 maintain a SpO2 between 90% to 94% for at least 30 min. Infants will also be given surfactant if their clinical status will deteriorate rapidly or will develop respiratory acidosis defined as a pCO2 more than 65 mmHg (8.5 kPa) and a pH less than 7.20, or with lung ultrasound scoring >8. A loading dose of intravenous caffeine citrate (20 mg/kg) will be given in the delivery room or immediately after admission to the NICU (within 2 hours of life) or in any case prior to surfactant administration, followed by a daily morning in-trave-nous dose of 5-10 mg/kg as required.

All neonates of both groups will receive preprocedural medications using intravenous atropine (10 µg/kg) in one minute followed by intravenous fentanyl: 0.5 µg/kg by pump infusion in no less than 5 minutes (possibly repeatable dose if satisfactory analgosedation is not obtained) or followed by in-travenous ketamine: 0.5 mg/kg in no less than one minute (possibly repeatable dose if satisfactory analgosedation is not obtained). Method of premedication will be documented in each participating centre.

IN-REC-SUR-E group infants after intubation, will receive HFOV starting at MAP 8 cmH2O; fre-quency 15 Hz, with volum guarantee (1.5-1.7 mL/kg). The I:E will be 1:1. An oxygenation guided lung recruitment procedure will be performed using stepwise increments then decrements in MAP. The starting MAP will be increased stepwise as long as SpO2 improves reducing the FiO2 keeping SpO2 within the target range (90-94 %) until the oxygenation no longer improves or the FiO2 is equal to or less than 0.25 (opening MAP). Next, the MAP will be reduced stepwise until the SpO2 deteriorates (closing MAP). After a second recruitment maneuver at the opening pressure, the opti-mal MAP will be set 2 cmH2O above the closing MAP. Then 200 mg/kg of poractant alfa (Chiesi Farmaceutici S.p.A., Parma, Italy) via a closed administration system will administrate. In-fants with sufficient respiratory drive will be extubated within 30 minutes after surfactant admin-istration start-ing nCPAP (7-9 cm H2O) or NIPPV.

LISA Group infants allocated will receive 200 mg/kg of poractant alfa (Chiesi Farmaceutici S.p.A., Parma, Italy) during nCPAP of 7-8 cmH2O. Surfactant will be administered over 0.5-3 min using the SurfCath™ tracheal instillation catheter (VYGON S.A. - Ecouen, France), or a 4- 6 F end-hole catheter. The infant's mouth will be closed. In cases of apnoea or bradycardia, positive pressure ven-tilation will be performed until recovery. After surfactant administration, CPAP (7-9 cm H2O) or NIPPV will be continued.

Transcutaneous PaCO2 will be recorded during surfactant administration in both the procedures (IN-REC-SUR-E and LISA), if available.

In nCPAP infants, the decision as to whether to begin bilevel positive airway pressure or NIPPV to prevent the need for re-intubation in infants of both groups will be up to the neonatologist on duty and will be considered in the final analysis. Infants in both groups who meet the CPAP/NIPPV fail-ure criteria again during the following 24 h will receive a second dose of surfactant (100 mg/kg of poractant alfa) according to the randomized group (IN-REC-SUR-E or LISA).

The indications for MV after IN-REC-SUR-E or LISA will be: Poor oxygenation with FiO2 of greater than 0.40 to maintain a SpO2 between 90% to 94% despite CPAP (7-9 cm H2O) or NIPPV; respiratory; apnoea, despite optimal noninvasive respiratory sup-port.

Primary outcome is a composite outcome of death or BPD at 36 weeks' postmenstrual age.

DATA COLLECTION AND MANAGMENT. A customized eCRF (eletronic Case Report Form) will be created for the study. Pseudo-anonimyzed study data will be collected and managed using REDCap electronic data capture tools hosted at Fondazione Policlinico Universitario A. Gemellli, IRCCS (https://redcap-irccs.policlinicogemelli.it/). All collected data will be obtained from the clini-cal records. All data above listed in "Primary out-come measure", "secondary outcome measure", and "Other collected data" sections. Adverse events, device deficiency and incidents will be rec-orded and reported to Manufacturer and the National Competent Authority as per applicable law.

Statistical analysis The investigators hypothesized that IN-REC-SUR-E technique for surfactant administration might increase the survival without BPD at 36 weeks of postmenstrual age in extremely preterm infants, respect to LISA approach, from 65 % to 80 %. The investigators based the 15 % difference estimate from the data of the German Neonatal Network (GNN) on the LISA approach, from the results of the OPTIMIST trial recently published and from updated data on the IN-REC-SUR-E technique of some Italian Centers that continued to use this strategy even after that the INRECSURE study had ended. The investigators calculated that 181 newborns must be enrolled in each group to detect this difference as statistically significant with 90 % power at 0.05 level. 381 patients will be randomly assigned to accommodate the risk of enrolling a 5% of patients judged not meeting inclusion criteria after randomization. Twins will be separately randomized. Analyses will be done according to the intention-to-treat and per-protocol principles, as suggested by CONSORT guidelines, with the primary outcome assessed in the in-ten-tion-to-treat population. The intention-to-treat population will include all participants assigned to study intervention, and the per-protocol population will include all participants who receive and complete the study intervention, and who met study criteria. For the primary outcome, a log-binomial regression model correcting for the stratification factors of gestational age and study centre will be used to estimate the adjusted relative risk (RR). Moreover, the absolute risk reduction and the number-needed-to-treat will be calculated. Statistical analyses will be done using Stata software, version 16. An interim-analysis for safety to evaluate the prespecified stopping rules will be done at 30 % of recruitment by an independent statistician, masked to the treatment allocation. The prespecified clinical and safety outcomes will be: in-hospital mortality, intraventricular haemor-rhage worse than grade 2 and pneumothorax. The data and safety monitoring board will have un-masked access to all data and will discuss the results of the interim analysis with the steer-ing com-mittee in a joint meeting. The steering committee will decide on the continuation of the trial and will report to the central ethics committee.

Duration of study: 3 years QUALITY CONTROL AND QUALITY ASSURANCE PROCEDURES Compliance to protocol Compliance will be defined as full adherence to protocol. Compliance with the protocol will be ensured by a number of procedures as: site set-up local principal investigators are required to participate in preparatory meetings in which details of study protocol, data collection, "IN-REC-SUR-E" and "LISA" procedures will be accurately discussed. All centers will receive de-tailed written instruction on web based data recording, and, to solve possible difficulties, it will be possible to contact the Clinical Trials Coordinating Center. Moreover, it has been ascertained that "IN-REC-SUR-E" and "LISA" procedures are followed similarly in all participating centers.

ELIGIBILITY:
Inclusion Criteria:

Infants satisfying the following inclusion criteria will be eligible to participate:

1. Born at 24+0-27+6 in a tertiary neonatal intensive care unit participating in the trial (and)
2. Breathing independently and sufficiently with only nasal CPAP or NIPPV for respiratory support (and)
3. Written parental consent has been obtained (and)
4. Failing nasal CPAP or NIPPV during the first 24 hours of life

Exclusion Criteria:

1. Severe birth asphyxia or a 5-minute Apgar score less than 3
2. Prior endotracheal intubation for resuscitation or insufficient respiratory drive
3. Prolonged (>21 days) premature rupture of membranes
4. Presence of major congenital abnormalities
5. Hydrops fetalis
6. Inherited disorders of metabolism

Ages: 24 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 381 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
A composite outcome of death or bronchopulmonary dysplasia (BPD) at 36 weeks' postmenstrual age | 36 weeks' postmenstrual age or death
  A composite outcome of death or bronchopulmonary dysplasia (BPD) at 36 weeks' postmenstrual age is the primary outcome because BPD represents the most severe respiratory morbidity of preterm infants and death is a competing risk. The diagnosis of BPD will be ascertained by a standardized test. Infants remaining on mechanical ventilation or CPAP at 36 weeks postmenstrual age, or those with a supplemental oxygen concentration ≥0.30 to obtain SpO2 between 90% to 94% will receive a BPD diagnosis without additional testing. Infants with a supplemental oxygen concentration < 0.30 to obtain SpO2 between 90% to 94% or those receiving high-flow nasal cannula therapy will undergo a timed stepwise reduction to room air without any flow. Those in whom the reduction will not be tolerated will receive a BPD diagnosis.

SECONDARY OUTCOMES:
BPD at 36 weeks' s postmenstrual age | 36 weeks' s postmenstrual age
  BPD at 36 weeks' s postmenstrual age
Death at 36 weeks' s postmenstrual age or before discharge | 36 weeks' s postmenstrual age or hospital stay
  Death at 36 weeks' s postmenstrual age or before discharge
SpO2/FiO2 at 3 days, 7 days, and thereafter every 7 days until 36 weeks postmenstrual age | 36 weeks postmenstrual age
  SpO2/FiO2 at 3 days, 7 days, and thereafter every 7 days until 36 weeks postmenstrual age
Severe intraventricular hemorrhage (grade 3 or 4 based on the Papile criteria) | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Severe intraventricular hemorrhage (grade 3 or 4 based on the Papile criteria) minimum: grade 3 maximum: grade 4 Grade 4 means a worse outcome
Occurrence of air leaks including pneumothorax or pulmonary interstitial emphysema before discharge | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Occurrence of air leaks including pneumothorax or pulmonary interstitial emphysema before discharge
Duration of invasive respiratory support | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Duration of invasive respiratory support
Duration of non-invasive respiratory support | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Duration of non-invasive respiratory support
Duration of oxygen therapy | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Duration of oxygen therapy
Rate of pulmonary Hemorrhage | First 72 hours of life
  Pulmonary hemorrhage
Rate of patent ductus arteriosus; haemodynamically significant (PDAhs) (i.e.requiring pharmacological treatment with ibuprofen/indomethacin/acetaminophen). | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Patent ductus arteriosus; haemodynamically significant (PDAhs) (i.e.requiring pharmacological treatment with ibuprofen/indomethacin/acetaminophen).
Percentage of infants receiving two or more doses of surfactant | First 72 hours of life
  Percentage of infants receiving two or more doses of surfactant
Incidence of periventricular leukomalacia (PVL) | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Incidence of periventricular leukomalacia (PVL)
Incidence of a grade 3 or above retinopathy of prematurity (ROP) | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Incidence of a grade 3 or above retinopathy of prematurity (ROP)
Incidence of any necrotizing enterocolitis (NEC) | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Incidence of any necrotizing enterocolitis (NEC)
Incidence of sepsis defined as a positive blood culture or suggestive clinical and laboratory findings leading to treatment with antibiotics for at least 7 days despite absence of a positive blood culture | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Incidence of sepsis defined as a positive blood culture or suggestive clinical and laboratory findings leading to treatment with antibiotics for at least 7 days despite absence of a positive blood culture
Total in-hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Total in-hospital stay
Rate of use of systemic postnatal steroids | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Use of systemic postnatal steroids
Neurodevelopmental outcomes via Bayley scales of infant development-III and respiratory function testing at 24 months of age. | 24 months of age
  Bayley III - Nancy Bayley (scales of infantand toddler development third edition) 45 minimum value and155 maximum value (higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Brix N, Sellmer A, Jensen MS, Pedersen LV, Henriksen TB. Predictors for an unsuccessful INtubation-SURfactant-Extubation procedure: a cohort study. BMC Pediatr. 2014 Jun 19;14:155. doi: 10.1186/1471-2431-14-155. PMID 24947477
- [Result] Svedenkrans J, Stoecklin B, Jones JG, Doherty DA, Pillow JJ. Physiology and Predictors of Impaired Gas Exchange in Infants with Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2019 Aug 15;200(4):471-480. doi: 10.1164/rccm.201810-2037OC. PMID 30789787
- [Result] Lakkundi A, Wright I, de Waal K. Transitional hemodynamics in preterm infants with a respiratory management strategy directed at avoidance of mechanical ventilation. Early Hum Dev. 2014 Aug;90(8):409-12. doi: 10.1016/j.earlhumdev.2014.04.017. Epub 2014 Jun 5. PMID 24951077
- [Result] Dani C, Corsini I, Bertini G, Fontanelli G, Pratesi S, Rubaltelli FF. The INSURE method in preterm infants of less than 30 weeks' gestation. J Matern Fetal Neonatal Med. 2010 Sep;23(9):1024-9. doi: 10.3109/14767050903572174. PMID 20180736
- [Result] Cherif A, Hachani C, Khrouf N. Risk factors of the failure of surfactant treatment by transient intubation during nasal continuous positive airway pressure in preterm infants. Am J Perinatol. 2008 Nov;25(10):647-52. doi: 10.1055/s-0028-1090590. Epub 2008 Oct 7. PMID 18841536
- [Result] Vento G, Ventura ML, Pastorino R, van Kaam AH, Carnielli V, Cools F, Dani C, Mosca F, Polglase G, Tagliabue P, Boni L, Cota F, Tana M, Tirone C, Aurilia C, Lio A, Costa S, D'Andrea V, Lucente M, Nigro G, Giordano L, Roma V, Villani PE, Fusco FP, Fasolato V, Colnaghi MR, Matassa PG, Vendettuoli V, Poggi C, Del Vecchio A, Petrillo F, Betta P, Mattia C, Garani G, Solinas A, Gitto E, Salvo V, Gargano G, Balestri E, Sandri F, Mescoli G, Martinelli S, Ilardi L, Ciarmoli E, Di Fabio S, Maranella E, Grassia C, Ausanio G, Rossi V, Motta A, Tina LG, Maiolo K, Nobile S, Messner H, Staffler A, Ferrero F, Stasi I, Pieragostini L, Mondello I, Haass C, Consigli C, Vedovato S, Grison A, Maffei G, Presta G, Perniola R, Vitaliti M, Re MP, De Curtis M, Cardilli V, Lago P, Tormena F, Orfeo L, Gizzi C, Massenzi L, Gazzolo D, Strozzi MCM, Bottino R, Pontiggia F, Berardi A, Guidotti I, Cacace C, Meli V, Quartulli L, Scorrano A, Casati A, Grappone L, Pillow JJ. Lung recruitment before surfactant administration in extremely preterm neonates with respiratory distress syndrome (IN-REC-SUR-E): a randomised, unblinded, controlled trial. Lancet Respir Med. 2021 Feb;9(2):159-166. doi: 10.1016/S2213-2600(20)30179-X. Epub 2020 Jul 17. PMID 32687801
- [Result] Kribs A. Minimally Invasive Surfactant Therapy and Noninvasive Respiratory Support. Clin Perinatol. 2016 Dec;43(4):755-771. doi: 10.1016/j.clp.2016.07.010. Epub 2016 Oct 14. PMID 27837757
- [Result] Bellos I, Fitrou G, Panza R, Pandita A. Comparative efficacy of methods for surfactant administration: a network meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2021 Sep;106(5):474-487. doi: 10.1136/archdischild-2020-319763. Epub 2021 Jan 15. PMID 33452218
- [Result] Nobile S, Bottoni A, Giordano L, Paladini A, Vento G. Critical appraisal of the evidence underpinning the efficacy of less invasive surfactant administration. Arch Dis Child Fetal Neonatal Ed. 2023 Jan;108(1):90-91. doi: 10.1136/archdischild-2021-323100. Epub 2021 Oct 16. No abstract available. PMID 34656993
- [Result] Janssen LC, Van Der Spil J, van Kaam AH, Dieleman JP, Andriessen P, Onland W, Niemarkt HJ. Minimally invasive surfactant therapy failure: risk factors and outcome. Arch Dis Child Fetal Neonatal Ed. 2019 Nov;104(6):F636-F642. doi: 10.1136/archdischild-2018-316258. Epub 2019 Apr 29. PMID 31036700
- [Result] Bellos I, Pandita A. SurE for surfactant: response to letter. Arch Dis Child Fetal Neonatal Ed. 2023 Jan;108(1):91-92. doi: 10.1136/archdischild-2021-323394. Epub 2021 Nov 29. No abstract available. PMID 34844986
- [Result] Finer NN, Katheria A. Recruitment: the best way to IN-SUR-E surfactant delivery? Lancet Respir Med. 2021 Feb;9(2):119-120. doi: 10.1016/S2213-2600(20)30242-3. Epub 2020 Jul 17. No abstract available. PMID 32687802
- [Result] Broglio K. Randomization in Clinical Trials: Permuted Blocks and Stratification. JAMA. 2018 Jun 5;319(21):2223-2224. doi: 10.1001/jama.2018.6360. No abstract available. PMID 29872845
- [Result] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Result] Aziz K, Lee HC, Escobedo MB, Hoover AV, Kamath-Rayne BD, Kapadia VS, Magid DJ, Niermeyer S, Schmolzer GM, Szyld E, Weiner GM, Wyckoff MH, Yamada NK, Zaichkin J. Part 5: Neonatal Resuscitation: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S524-S550. doi: 10.1161/CIR.0000000000000902. Epub 2020 Oct 21. No abstract available. PMID 33081528
- [Result] De Jaegere A, van Veenendaal MB, Michiels A, van Kaam AH. Lung recruitment using oxygenation during open lung high-frequency ventilation in preterm infants. Am J Respir Crit Care Med. 2006 Sep 15;174(6):639-45. doi: 10.1164/rccm.200603-351OC. Epub 2006 Jun 8. PMID 16763218
- [Result] Buzzella B, Claure N, D'Ugard C, Bancalari E. A randomized controlled trial of two nasal continuous positive airway pressure levels after extubation in preterm infants. J Pediatr. 2014 Jan;164(1):46-51. doi: 10.1016/j.jpeds.2013.08.040. Epub 2013 Oct 1. PMID 24094879
- [Result] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Result] Walsh MC, Szefler S, Davis J, Allen M, Van Marter L, Abman S, Blackmon L, Jobe A. Summary proceedings from the bronchopulmonary dysplasia group. Pediatrics. 2006 Mar;117(3 Pt 2):S52-6. doi: 10.1542/peds.2005-0620I. PMID 16777823
- [Result] Nobile S, Marchionni P, Gidiucci C, Correani A, Palazzi ML, Spagnoli C, Rondina C; Marche Neonatal Network; Carnielli VP. Oxygen saturation/FIO2 ratio at 36 weeks' PMA in 1005 preterm infants: Effect of gestational age and early respiratory disease patterns. Pediatr Pulmonol. 2019 May;54(5):637-643. doi: 10.1002/ppul.24265. Epub 2019 Jan 27. PMID 30688034
- [Result] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Result] de Vries LS, Eken P, Dubowitz LM. The spectrum of leukomalacia using cranial ultrasound. Behav Brain Res. 1992 Jul 31;49(1):1-6. doi: 10.1016/s0166-4328(05)80189-5. PMID 1388792
- [Result] International Committee for the Classification of Retinopathy of Prematurity. The International Classification of Retinopathy of Prematurity revisited. Arch Ophthalmol. 2005 Jul;123(7):991-9. doi: 10.1001/archopht.123.7.991. PMID 16009843
- [Result] Bell MJ, Ternberg JL, Feigin RD, Keating JP, Marshall R, Barton L, Brotherton T. Neonatal necrotizing enterocolitis. Therapeutic decisions based upon clinical staging. Ann Surg. 1978 Jan;187(1):1-7. doi: 10.1097/00000658-197801000-00001. PMID 413500
- [Result] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Result] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Result] Dargaville PA, Kamlin COF, Orsini F, Wang X, De Paoli AG, Kanmaz Kutman HG, Cetinkaya M, Kornhauser-Cerar L, Derrick M, Ozkan H, Hulzebos CV, Schmolzer GM, Aiyappan A, Lemyre B, Kuo S, Rajadurai VS, O'Shea J, Biniwale M, Ramanathan R, Kushnir A, Bader D, Thomas MR, Chakraborty M, Buksh MJ, Bhatia R, Sullivan CL, Shinwell ES, Dyson A, Barker DP, Kugelman A, Donovan TJ, Tauscher MK, Murthy V, Ali SKM, Yossuck P, Clark HW, Soll RF, Carlin JB, Davis PG; OPTIMIST-A Trial Investigators. Effect of Minimally Invasive Surfactant Therapy vs Sham Treatment on Death or Bronchopulmonary Dysplasia in Preterm Infants With Respiratory Distress Syndrome: The OPTIMIST-A Randomized Clinical Trial. JAMA. 2021 Dec 28;326(24):2478-2487. doi: 10.1001/jama.2021.21892. PMID 34902013
- [Result] Ranganathan P, Pramesh CS, Aggarwal R. Common pitfalls in statistical analysis: Intention-to-treat versus per-protocol analysis. Perspect Clin Res. 2016 Jul-Sep;7(3):144-6. doi: 10.4103/2229-3485.184823. PMID 27453832
- [Derived] Vento G, Paladini A, Aurilia C, Ozdemir SA, Carnielli VP, Cools F, Costa S, Cota F, Dani C, Davis PG, Fattore S, Fe C, Finer N, Fusco FP, Gizzi C, Herting E, Jian M, Lio A, Lista G, Mosca F, Nobile S, Perri A, Picone S, Pillow JJ, Polglase G, Pasciuto T, Pastorino R, Tana M, Tingay D, Tirone C, van Kaam AH, Ventura ML, Aceti A, Agosti M, Alighieri G, Ancora G, Angileri V, Ausanio G, Aversa S, Balestri E, Baraldi E, Barbini MC, Barone C, Beghini R, Bellan C, Berardi A, Bernardo I, Betta P, Binotti M, Bizzarri B, Borgarello G, Borgione S, Borrelli A, Bottino R, Bracaglia G, Bresesti I, Burattini I, Cacace C, Calzolari F, Campagnoli MF, Capasso L, Capozza M, Capretti MG, Caravetta J, Carbonara C, Cardilli V, Carta M, Castoldi F, Castronovo A, Cavalleri E, Cavigioli F, Cecchi S, Chierici V, Cimino C, Cocca F, Cocca C, Cogo P, Coma M, Comito V, Condo V, Consigli C, Conti R, Corradi M, Corsello G, Corvaglia LT, Costa A, Coscia A, Cresi F, Crispino F, D'Amico P, De Cosmo L, De Maio C, Del Campo G, Di Credico S, Di Fabio S, Di Nicola P, Di Paolo A, Di Valerio S, Distilo A, Duca V, Falcone A, Falsaperla R, Fasolato VA, Fatuzzo V, Favini F, Ferrarello MP, Ferrari S, Nastro FF, Forcellini CA, Fracchiolla A, Gabriele A, Galdo F, Gallini F, Gangemi A, Gargano G, Gazzolo D, Gentile MP, Ghirardello S, Giardina F, Giordano L, Gitto E, Giuffre M, Grappone L, Grasso F, Greco I, Grison A, Guglielmino R, Guidotti I, Guzzo I, La Forgia N, La Placa S, La Torre G, Lago P, Lanciotti L, Lavizzari A, Leo F, Leonardi V, Lestingi D, Li J, Liberatore P, Lodin D, Lubrano R, Lucente M, Luciani S, Luvara D, Maffei G, Maggio A, Maggio L, Maiolo K, Malaigia L, Mangili G, Manna A, Maranella E, Marciano A, Marcozzi P, Marletta M, Marseglia L, Martinelli D, Martinelli S, Massari S, Massenzi L, Matina F, Mattia L, Mescoli G, Migliore IV, Minghetti D, Mondello I, Montano S, Morandi G, Mores N, Morreale S, Morselli I, Motta M, Napolitano M, Nardo D, Nicolardi A, Nider S, Nigro G, Nuccio M, Orfeo L, Ottaviano C, Paganin P, Palamides S, Palatta S, Paolillo P, Pappalardo MG, Pasta E, Patti L, Paviotti G, Perniola R, Perotti G, Perrone S, Petrillo F, Piazza MS, Piccirillo A, Pierro M, Piga E, Pingitore GA, Pisu S, Pittini C, Pontiggia F, Pontrelli G, Primavera A, Proto A, Quartulli L, Raimondi F, Ramenghi L, Rapsomaniki M, Ricotti A, Rigotti C, Rinaldi M, Risso FM, Roma E, Romanini E, Romano V, Rosati E, Rosella V, Rulli I, Salvo V, Sanfilippo C, Sannia A, Saporito A, Sauna A, Scapillati E, Schettini F, Scorrano A, Mantelli SS, Sepporta V, Sindico P, Solinas A, Sorrentino E, Spaggiari E, Staffler A, Stella M, Termini D, Terrin G, Testa A, Tina G, Tirantello M, Tomasini B, Tormena F, Travan L, Trevisanuto D, Tuling G, Tulino V, Valenzano L, Vedovato S, Vendramin S, Villani PE, Viola S, Viola V, Vitaliti G, Vitaliti M, Wanker P, Yang Y, Zanetta S, Zannin E. Comparison of "IN-REC-SUR-E" and LISA in preterm neonates with respiratory distress syndrome: a randomized controlled trial (IN-REC-LISA trial). Trials. 2024 Jul 2;25(1):433. doi: 10.1186/s13063-024-08240-4. PMID 38956676